CLINICAL TRIAL: NCT04619251
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses and Multiple Oral Doses of BI 1323495 Versus Placebo in Healthy Male Japanese Subjects Genotyped as Poor and Extensive Metabolizers of UGT2B17 (Single-blind, Randomised, Placebo-controlled [Within Dose Groups] Trial), Including an Investigation of Drug-drug Interaction With Itraconazole in Healthy Male Subjects Genotyped as Poor Metabolizers of UGT2B17 (an Open-label, Two-period, Fixed Sequence Trial)
Brief Title: A Study in Healthy Japanese Men to Test How Different Doses of BI 1323495 Are Tolerated and How Itraconazole Influences the Amount of BI 1323495 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1405-0003
Record Dates: First submitted 2020-10-28; First posted 2020-11-06 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- SRD part: PM Subjects, BI1323495 10mg (Experimental): Participants were administered on Day 1 a single oral dose of 10 milligram (mg) of BI 1323495 film-coated tablet together with about 240 milliliter (mL) of water. A standardized meal was served 30 minutes (min) before drug administration. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 1323495
- SRD part: PM Subjects, BI1323495 30mg (Experimental): Participants were administered on Day 1 a single oral dose of 30 milligram (mg) of BI 1323495 film-coated tablets together with about 240 milliliter (mL) of water. A standardized meal was served 30 minutes (min) before drug administration.
  One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 1323495
- SRD part: PM Subjects, BI1323495 100mg (Experimental): Participants were administered on Day 1 a single oral dose of 100 milligram (mg) of BI 1323495 film-coated tablets together with about 240 milliliter (mL) of water. A standardized meal was served 30 minutes (min) before drug administration. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 1323495
- SRD part: EM Subjects, BI1323495 30mg (Experimental): Participants were administered on Day 1 a single oral dose of 30 milligram (mg) of BI 1323495 film-coated tablets together with about 240 milliliter (mL) of water. A standardized meal was served 30 minutes (min) before drug administration. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 1323495
- SRD part: EM Subjects, BI1323495 70mg (Experimental): Participants were administered on Day 1 a single oral dose of 70 milligram (mg) of BI 1323495 film-coated tablets together with about 240 milliliter (mL) of water. A standardized meal was served 30 minutes (min) before drug administration. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 1323495
- SRD part: EM Subjects, BI1323495 150mg (Experimental): Participants were administered on Day 1 a single oral dose of 150 milligram (mg) of BI 1323495 film-coated tablets together with about 240 milliliter (mL) of water. A standardized meal was served 30 minutes (min) before drug administration. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 1323495
- SRD part: Placebo (Placebo Comparator): This arm comprises all placebo treated participants in trial part SRD, regardless of the dose group in which they were treated. Participants were randomized within each dose group in a 3:1 ratio (test treatment to placebo).
  Participants were administered on Day 1 a single oral dose of placebo film-coated tablet(s) together with about 240 milliliter (mL) of water. A standardized meal was served 30 minutes (min) before drug administration. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: Placebo
- MD part: PM Subjects, BI1323495 30mg BID (Experimental): Participants were administered from Day 1 to Day 10 two times per day (bid) an oral dose of 30 milligram (mg) of BI 1323495 film-coated tablets together with about 240 milliliter (mL) of water, At Day 11 participants were administered only a single dose in the morning. Participants took a normal caloric meal 30 minutes (min) before drug administration. Subjects fasted for 4 hours (h) after intake of morning dose. Morning and evening dose were taken with a 12 h time interval approximately at the same time each day during the treatment phase. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 1323495
- MD part: PM Subjects, BI1323495 60mg QD (Experimental): Participants were administered from Day 1 to Day 11 one time per day (qd) an oral dose of 60 milligram (mg) of BI 1323495 film-coated tablets together with about 240 milliliter (mL) of water. Participants took a normal caloric meal 30 minutes (min) before drug administration. Subjects fasted for 4 hours (h) after intake of morning dose. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: BI 1323495
- MD part: Placebo (Placebo Comparator): This arm comprises all placebo treated participants in trial part MD, regardless of the dose group in which they were treated. Participants were randomized within each dose group in a 3:1 ratio (test treatment to placebo). Participants were administered from Day 1 to Day 11 one time per day (qd) an oral dose of placebo film-coated tablets or two times per day (bid) an oral dose of placebo together with about 240 milliliter (mL) of water. Participants took a normal caloric meal 30 minutes (min) before drug administration. Subjects fasted for 4 hours (h) after intake of morning dose. One authorized employee of the trial site was witness of the administration of the trial medication.
  Interventions: Drug: Placebo
- DDI part: PM Subjects, BI1323495 / BI1323495+ Itraconazole (Experimental): * Period 1: Participants were administered the reference treatment (R) which consisted of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 together with about 240 milliliter (mL) of water on Day 1 of Period 1. One authorized employee of the trial site was witness of the administration of the trial medication.
  * Period 2: Participants were administered the test treatment (T) which consisted of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 with about 240 milliliter (mL) of water on Day 1 of Period 2, together with multiple oral doses of 200 mg itraconazole from Day -3 to Day 7, in total 10 doses, as oral solution formulation. One authorized employee of the trial site was witness of the administration of the trial medication.
  Administration of BI 1323495 in treatment R and T were separated by at least 11 days.
  Interventions: Drug: BI 1323495; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 1323495 — BI 1323495
  Arms: DDI part: PM Subjects, BI1323495 / BI1323495+ Itraconazole; MD part: PM Subjects, BI1323495 30mg BID; MD part: PM Subjects, BI1323495 60mg QD; SRD part: EM Subjects, BI1323495 150mg; SRD part: EM Subjects, BI1323495 30mg; SRD part: EM Subjects, BI1323495 70mg; SRD part: PM Subjects, BI1323495 100mg; SRD part: PM Subjects, BI1323495 10mg; SRD part: PM Subjects, BI1323495 30mg
Drug: Placebo — Placebo
  Arms: MD part: Placebo; SRD part: Placebo
Drug: Itraconazole — Itraconazole
  Arms: DDI part: PM Subjects, BI1323495 / BI1323495+ Itraconazole

SUMMARY:
The main objective of the single-rising dose (SRD) part and the multiple rising dose (MD) part is to investigate safety, tolerability, pharmacokinetics and pharmacodynamics (for MD part only) following single rising doses and multiple oral doses of BI 1323495 in healthy male Japanese subjects genotyped as poor metabolizers (PM) and extensive metabolizers (EM) of UGT2B17.

The main objective of the drug-drug interaction (DDI) part is to investigate the relative bioavailability of a single oral dose of BI 1323495 when given alone (treatment R) or in combination with itraconazole (treatment T) in healthy male subjects genotyped as PM of UGT2B17.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history, including a medical examination, vital signs (BP, PR), 12- lead ECG, and clinical laboratory tests
* Japanese ethnicity, according to the following criteria:

  --born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 20 to 45 years (inclusive) at screening
* BMI of 18.5 to 25.0 kg/m2 (inclusive) at screening
* Signed and dated written informed consent prior to admission to the trial, in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who agree to minimize the risk of making their partner pregnant by fulfilling any of the following criteria starting from the first administration of trial medication until 90 days after last administration of trial medication
* Use of adequate contraception, any of the following methods plus condom: intrauterine device, combined oral contraceptives that started at least 2 months prior to the first drug administration.
* Vasectomized (vasectomy at least 1 year prior to enrolment)
* Surgical sterilization (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner
* Subjects genotyped as UGT2B17 poor metabolizers, i.e. carrying allele of UGT2B17 gene (*2/*2) (DDI part only)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 40 to 90 mmHg, or pulse rate outside the range of 40 to 99 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two part clinical trial, the first part was single rising dose (SRD) and multiple dose (MD), the second part evaluates drug-drug interaction (DDI) with itraconazole. The study was performed in healthy Japanese men genotyped as poor metabolizers (PM) or as extensive metabolizers (EM) to test how different doses of BI 1323495 are tolerated and how itraconazole influences the amount of BI 1323495 in the blood.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. Administrations of BI 1323495 was separated by a wash-out phase of at least 11 days.
Period: Period 1
Arm/Group | SRD Part: PM Subjects, BI1323495 10mg | SRD Part: PM Subjects, BI1323495 30mg | SRD Part: PM Subjects, BI1323495 100mg | SRD Part: EM Subjects, BI1323495 30mg | SRD Part: EM Subjects, BI1323495 70mg | SRD Part: EM Subjects, BI1323495 150mg | SRD Part: Placebo | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD | MD Part: Placebo | DDI Part: PM Subjects, BI1323495 / BI1323495+ Itraconazole
Started | 6 | 6 | 6 | 3 | 3 | 3 | 9 | 9 | 9 | 6 | 14
Completed | 6 | 6 | 6 | 3 | 3 | 3 | 9 | 9 | 9 | 6 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | SRD Part: PM Subjects, BI1323495 10mg | SRD Part: PM Subjects, BI1323495 30mg | SRD Part: PM Subjects, BI1323495 100mg | SRD Part: EM Subjects, BI1323495 30mg | SRD Part: EM Subjects, BI1323495 70mg | SRD Part: EM Subjects, BI1323495 150mg | SRD Part: Placebo | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD | MD Part: Placebo | DDI Part: PM Subjects, BI1323495 / BI1323495+ Itraconazole
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who were randomised (SRD and MD part) / allocated (DDI part) and treated with at least one dose of trial drug. The treatment assignment will be determined based on the first treatment the subjects received. The treated set will be used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | SRD Part: PM Subjects, BI1323495 10mg | SRD Part: PM Subjects, BI1323495 30mg | SRD Part: PM Subjects, BI1323495 100mg | SRD Part: EM Subjects, BI1323495 30mg | SRD Part: EM Subjects, BI1323495 70mg | SRD Part: EM Subjects, BI1323495 150mg | SRD Part: Placebo | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD | MD Part: Placebo | DDI Part: PM Subjects, BI1323495 / BI1323495+ Itraconazole | Total
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 3 | 3 | 9 | 9 | 9 | 6 | 14 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.3 (3.8) | 32.5 (10.3) | 33.5 (7.6) | 24.7 (3.1) | 33.0 (4.6) | 29.3 (5.5) | 29.3 (7.0) | 32.3 (5.6) | 28.6 (4.6) | 30.0 (6.5) | 30.4 (7.2) | 30.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 3 | 3 | 3 | 9 | 9 | 9 | 6 | 14 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 3 | 3 | 3 | 9 | 9 | 9 | 6 | 14 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 3 | 3 | 3 | 9 | 9 | 9 | 6 | 14 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: SRD and MD Part: Number of Participants With Drug-related Adverse Events (AEs)
Description: Number of participants with drug-related adverse events (AEs) is reported for Single rising dose (SRD) and Multiple dose (MD) parts is reported.
Time Frame: Up to 7 days (for SRD part), up to 17 days (for MD part).
Population: Treated set (TS): The treated set includes all subjects who were randomised (SRD and MD part) and treated with at least one dose of trial drug. As pre-specified in the protocol this endpoint only includes the SRD and MD part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SRD Part: PM Subjects, BI1323495 10mg | SRD Part: PM Subjects, BI1323495 30mg | SRD Part: PM Subjects, BI1323495 100mg | SRD Part: EM Subjects, BI1323495 30mg | SRD Part: EM Subjects, BI1323495 70mg | SRD Part: EM Subjects, BI1323495 150mg | SRD Part: Placebo | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD | MD Part: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 3 | 3 | 9 | 9 | 9 | 6
Participants | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 1

2. Primary Outcome: DDI Part: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: The area under the concentration-time curve of BI 1323495 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported. The statistical model used for the analysis of this endpoint was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: subject and treatment. The effect 'subject' was considered as random, whereas the effect 'treatment' was considered as fixed. These quantities were then back-transformed to the original scale.
Time Frame: Within 3 hours (h) before and 20min, 40min, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h, 24h, 34h, 47h, 71h, 95h, 119h, 143h, and 167h after start of BI 1323495 administration on both periods (1 and 2).
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one primary or secondary PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only subjects with non-missing values were included.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanomol / liter (h*nmol/L)
Groups:
- DDI Part: BI1323495, Period 1: Participants were administered the reference treatment (R) which consisted of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 together with about 240 milliliter (mL) of water on Day 1 of Period 1. One authorized employee of the trial site was witness of the administration of the trial medication.
  Administration of BI 1323495 in treatment R and T were separated by at least 11 days.
- DDI Part: BI1323495+Itraconazole, Period 2: Participants were administered the test treatment (T) which consisted of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 with about 240 milliliter (mL) of water on Day 1 of Period 2, together with multiple oral doses of 200 mg itraconazole from Day -3 to Day 7, in total 10 doses, as oral solution formulation. One authorized employee of the trial site was witness of the administration of the trial medication.
  Administration of BI 1323495 in treatment R and T were separated by at least 11 days.
Arm/Group | DDI Part: BI1323495, Period 1 | DDI Part: BI1323495+Itraconazole, Period 2
Number analyzed (Participants) | 13 | 14
hour * nanomol / liter (h*nmol/L) | 757.8 (NA) — The standard error is actually the geometric standard error and is equal to 1.054. | 2558.3 (NA) — The standard error is actually the geometric standard error and is equal to 1.052
Statistical Analysis 1: Comparison: DDI Part: BI1323495, Period 1 vs DDI Part: BI1323495+Itraconazole, Period 2; The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: subject and treatment. The effect 'subject' was considered as random, whereas the effect 'treatment' was considered as fixed. These quantities were then back-transformed to the original scale; Test type: Other — Since the main focus is on estimation and not testing, a formal hypothesis test and associated acceptance range is not specified; Geometric Least Squares Mean ratio (%) = 337.6, 90% CI 2-sided [302.8 to 376.4] — Geometric Least Squares Mean ratio was estimated by the ratios of the geometric means (T/R). Intra-individual geometric coefficient variation (gCV %) =15.9

3. Primary Outcome: DDI Part: Maximum Measured Concentration of BI 1323495 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1323495 in plasma is reported. The statistical model used for the analysis of this endpoint was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: subject and treatment. The effect 'subject' was considered as random, whereas the effect 'treatment' was considered as fixed. These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one primary or secondary PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomol / liter (nmol/L)
Groups:
- DDI Part: BI1323495+ Itraconazole, Period 2: Participants were administered the test treatment (T) which consisted of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 with about 240 milliliter (mL) of water on Day 1 of Period 2, together with multiple oral doses of 200 mg itraconazole from Day -3 to Day 7, in total 10 doses, as oral solution formulation. One authorized employee of the trial site was witness of the administration of the trial medication, Administration of BI 1323495 in treatment R and T were separated by at least 11 days.
Arm/Group | DDI Part: BI1323495, Period 1 | DDI Part: BI1323495+ Itraconazole, Period 2
Number analyzed (Participants) | 14 | 14
nanomol / liter (nmol/L) | 81.2 (NA) — The standard error is actually the geometric standard error and is equal to 1.072. | 149.7 (NA) — The standard error is actually the geometric standard error and is equal to 1.072.
Statistical Analysis 1: Comparison: DDI Part: BI1323495, Period 1 vs DDI Part: BI1323495+ Itraconazole, Period 2; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; Geometric Least Squares Mean ratio (%) = 184.4, 90% CI 2-sided [156.0 to 218.0] — Geometric Least Squares Mean ratio was estimated by the ratios of the geometric means (T/R). Intra-individual geometric coefficient variation (gCV %) =26.4

4. Secondary Outcome: DDI Part: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: The area under the concentration-time curve BI 1323495 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported. The statistical model used for the analysis of this endpoint was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: subject and treatment. The effect 'subject' was considered as random, whereas the effect 'treatment' was considered as fixed. These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanomol / liter (h*nmol/L)
Groups:
- DDI Part: BI1323495+ Itraconazole, Period 2: Participants were administered the test treatment (T) which consisted of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 with about 240 milliliter (mL) of water on Day 1 of Period 2, together with multiple oral doses of 200 mg itraconazole from Day -3 to Day 7, in total 10 doses, as oral solution formulation. One authorized employee of the trial site was witness of the administration of the trial medication.
  Administration of BI 1323495 in treatment R and T were separated by at least 11 days.
Arm/Group | DDI Part: BI1323495, Period 1 | DDI Part: BI1323495+ Itraconazole, Period 2
Number analyzed (Participants) | 14 | 14
hour * nanomol / liter (h*nmol/L) | 704.5 (NA) — The standard error is actually the geometric standard error and is equal to 1.056. | 2513.8 (NA) — The standard error is actually the geometric standard error and is equal to 1.056.
Statistical Analysis 1: Comparison: DDI Part: BI1323495, Period 1 vs DDI Part: BI1323495+ Itraconazole, Period 2; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; Geometric Least Squares Mean ratio (%) = 356.8, 90% CI 2-sided [315.7 to 403.2] — Geometric Least Squares Mean ratio was estimated by the ratios of the geometric means (T/R). Intra-individual geometric coefficient variation (gCV %) =18.4

5. Secondary Outcome: SRD Part: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: The area under the concentration-time curve of BI 1323495 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
Time Frame: Within 3 hours (h) before and 20min, 40min, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h, 24h, 34h, 48h, 72h, 96h after start of BI 1323495 administration. Additionally only in the PM group: at 120h, 144h, and 168h.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomol / liter (h*nmol/L)
Arm/Group | SRD Part: PM Subjects, BI1323495 10mg | SRD Part: PM Subjects, BI1323495 30mg | SRD Part: PM Subjects, BI1323495 100mg | SRD Part: EM Subjects, BI1323495 30mg | SRD Part: EM Subjects, BI1323495 70mg | SRD Part: EM Subjects, BI1323495 150mg
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 3 | 3
hour * nanomol / liter (h*nmol/L) | 776 (9.14) | 2140 (25.7) | 6700 (13.9) | 715 (55.0) | 4040 (25.6) | 3550 (42.2)

6. Secondary Outcome: SRD Part: Maximum Measured Concentration of BI 1323495 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1323495 in plasma (Cmax) is reported.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol / liter (nmol/L)
Arm/Group | SRD Part: PM Subjects, BI1323495 10mg | SRD Part: PM Subjects, BI1323495 30mg | SRD Part: PM Subjects, BI1323495 100mg | SRD Part: EM Subjects, BI1323495 30mg | SRD Part: EM Subjects, BI1323495 70mg | SRD Part: EM Subjects, BI1323495 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 3 | 3
nanomol / liter (nmol/L) | 105 (18.0) | 276 (22.1) | 643 (9.15) | 86.9 (37.0) | 196 (8.72) | 230 (54.9)

7. Secondary Outcome: MD Part: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over the Time Interval of 12 h After Administration of the First Dose (AUC0-12)
Description: The area under the concentration-time curve of BI 1323495 in plasma over the time interval of 12 h after administration of the first dose (AUC0-12) is reported.
Time Frame: Within 3 hours (h) before and 20min, 40min, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h, after start of first dose BI 1323495 administration.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomol / liter (h*nmol/L)
Arm/Group | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD
Number analyzed (Participants) | 9 | 9
hour * nanomol / liter (h*nmol/L) | 1520 (15.4) | 2350 (15.1)

8. Secondary Outcome: MD Part: Maximum Measured Concentration of BI 1323495 in Plasma (Cmax) After First Dose
Description: Maximum measured concentration of BI 1323495 in plasma (Cmax) after first dose is reported.
Time Frame: as for outcome 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol / liter (nmol/L)
Arm/Group | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD
Number analyzed (Participants) | 9 | 9
nanomol / liter (nmol/L) | 303 (14.0) | 431 (15.2)

9. Secondary Outcome: MD Part: Area Under the Concentration-time Curve of BI 1323495 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss) After Last Dose Administration.
Description: Area under the concentration-time curve of BI 1323495 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) after last dose administration is reported. T for 30 mg bid is 12h, for 60 mg qd is 24h.
Time Frame: Within 15 minutes (min) before and 20min, 40min, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h and 24h (only for the 60mg qd administration) after last dose administration.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomol / liter (h*nmol/L)
Arm/Group | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD
Number analyzed (Participants) | 9 | 9
hour * nanomol / liter (h*nmol/L) | 2600 (20.0) | 4770 (17.0)

10. Secondary Outcome: MD Part: Maximum Measured Concentration of BI 1323495 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: Maximum measured concentration of BI 1323495 in plasma (Cmax,ss) at steady state over a uniform dosing interval τ is reported. T for 30 mg bid is 12h, for 60 mg qd is 24h.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol / liter (nmol/L)
Arm/Group | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD
Number analyzed (Participants) | 9 | 9
nanomol / liter (nmol/L) | 417 (17.1) | 570 (19.7)

ADVERSE EVENTS:
Time Frame: Up to 7 days for the SRD part, Up to 17 days for the MD part, Up to 7 days for the DDI-BI 1323495, Up to 3 days for the DDI-itraconazole, Up to 15 days for the DDI-BI1323495.+ itraconazole.
Description: Treated set (TS): The treated set includes all subjects who were randomized (SRD and MD part) / allocated (DDI part) and treated with at least one dose of trial drug.
  The Adverse Event assessment was reported for the DDI part: BI 1323495 (Period 1), subsequently the Itraconazole treatment and, for BI 1323495+Itraconazole treatment separately.
Groups:
- DDI Part: PM Subjects, BI1323495: During period 1, participants were administered the reference treatment (R) which consisted of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 together with about 240 milliliter (mL) of water on Day 1 of Period 1. One authorized employee of the trial site was witness of the administration of the trial medication. Administration of BI 1323495 in treatment R and T were separated by at least 11 days.
- DDI Part: PM Subjects, Itraconazole: During period 2, participants were administered the test treatment (T) which consisted of multiple oral doses of 200 mg itraconazole from Day -3 to Day 7, in total 10 doses, as oral solution formulation, together with of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 with about 240 milliliter (mL) of water on Day 1 of Period 2. Administration of BI 1323495 in treatment R and T were separated by at least 11 days.
- DDI Part: PM Subjects, BI1323495+ Itraconazole: During period 2, participants were administered the test treatment (T) which consisted of a single oral dose of 10 milligram (mg) film-coated tablet of BI 1323495 with about 240 milliliter (mL) of water on Day 1 of Period 2, together with multiple oral doses of 200 mg itraconazole from Day -3 to Day 7, in total 10 doses, as oral solution formulation. Administration of BI 1323495 in treatment R and T were separated by at least 11 days.
Arm/Group | SRD Part: Placebo | MD Part: Placebo | SRD Part: PM Subjects, BI1323495 10mg | SRD Part: PM Subjects, BI1323495 30mg | SRD Part: PM Subjects, BI1323495 100mg | SRD Part: EM Subjects, BI1323495 30mg | SRD Part: EM Subjects, BI1323495 70mg | SRD Part: EM Subjects, BI1323495 150mg | MD Part: PM Subjects, BI1323495 30mg BID | MD Part: PM Subjects, BI1323495 60mg QD | DDI Part: PM Subjects, BI1323495 | DDI Part: PM Subjects, Itraconazole | DDI Part: PM Subjects, BI1323495+ Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/3 | 0/3 | 0/9 | 0/9 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/3 | 0/3 | 0/9 | 0/9 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/9 | 1/6 | 1/6 | 2/6 | 4/6 | 2/3 | 1/3 | 0/3 | 2/9 | 4/9 | 4/14 | 1/14 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SRD Part: Placebo (N=9) | MD Part: Placebo (N=6) | SRD Part: PM Subjects, BI1323495 10mg (N=6) | SRD Part: PM Subjects, BI1323495 30mg (N=6) | SRD Part: PM Subjects, BI1323495 100mg (N=6) | SRD Part: EM Subjects, BI1323495 30mg (N=3) | SRD Part: EM Subjects, BI1323495 70mg (N=3) | SRD Part: EM Subjects, BI1323495 150mg (N=3) | MD Part: PM Subjects, BI1323495 30mg BID (N=9) | MD Part: PM Subjects, BI1323495 60mg QD (N=9) | DDI Part: PM Subjects, BI1323495 (N=14) | DDI Part: PM Subjects, Itraconazole (N=14) | DDI Part: PM Subjects, BI1323495+ Itraconazole (N=14)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 1 | 4 | 4 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT04619251/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT04619251/SAP_001.pdf